CLINICAL TRIAL: NCT02062398
Title: Safety and Performance of the BlueWind Medical Reprieve System for the Treatment of Patients With Peripheral Neuropathic Pain (PNP)
Brief Title: BlueWind Medical Reprieve System for the Treatment of PNP
Acronym: PNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BlueWind Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-02-001
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2018-11

CONDITIONS: Peripheral Neuropathy
Keywords: PNP; Stimulation; Peripheral neurostimulation
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The Reprieve system implantation (Experimental): The Reprieve implant will be implanted for eligible patients. Implant parameter settings will be set according to patient's sensations.
  Interventions: Device: The Reprieve System

INTERVENTIONS:
Device: The Reprieve System — BlueWind Medical neurostimulator for the treatment of neuropathic pain

SUMMARY:
The current study will evaluate the safety and performance of the BlueWind Medical Reprieve System for the treatment of Chronic Painful Peripheral Neuropathy.

DETAILED DESCRIPTION:
The BlueWind Reprieve system is a neurostimulator consisting of an Implant and external components.

The system is intended for home care use. The chronic pain treatment is achieved by an electrical stimulation of peripheral nerve fibers. The stimulation is set so that it generates paresthesia in the stimulated area (e.g. foot), reducing the pain sensation and improving the quality of life for the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Male or female aged 18 - 80.
3. Patient agrees to attend all follow-up evaluations and is willing to completely and accurately fill out pain questionnaires.
4. Diagnosis of chronic neuropathic pain due to peripheral neuropathy.
5. Documented pain attributed to neuropathy for at least 6 months.
6. Pain intensity with an average daily VAS score of at least 6, demonstrated by 2-3 ratings per day across 7 days.
7. Patient refractory to conservative treatments including pain medication, for at least 6 months.
8. Stable pain medication for at least 4 weeks prior to study enrollment.

Exclusion Criteria:

1. Previous participation in another study with any investigational drug or device within the past 90 days.
2. Any active implant (cardiac or other).
3. Any metal implant in the area of BlueWind device implantation site.
4. Current pregnancy or attempting to get pregnant (female patient).
5. Any clinically significant neurologic disorders (except PNP).
6. Any clinically significant or unstable medical or psychiatric condition that would affect the patient's ability to participate in the study.
7. Patients with severe or unstable cardiovascular, pulmonary, gastrointestinal, hematological, hepatic, renal or endocrine diseases.
8. Severe peripheral vascular disease that may cause intermittent claudication or ischemic ulcers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Pierre Van Buyten, MD, Principal Investigator — Sint-Niklaas hospital
Locations (4):
- Belgium (2):
  - AZ Sint-Jan Brugge - Oostende AV, Bruges
  - AZ Sint-Niklaas Hospital, Sint-Niklaas
- Poland (2):
  - 10 Military Clinical Hospital, Bydgoszcz
  - CenterMed Kraków Sp.z o.o., Krakow

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | The Reprieve System Implantation
Started | 13
Completed | 12
Not Completed | 1
Not completed — Implant removal | 1

BASELINE CHARACTERISTICS:
Arm/Group | The Reprieve System Implantation
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 59.7 [40 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
pain measurement using Visual Analogue Scale [Mean (Standard Deviation); unit: units on a scale] — Visual Analogue Scale for Pain 0 (no pain) - 10 (max pain) higher values represent a worse outcome
  units on a scale | 7.58 (1.11)

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of System and/or Procedure Related Serious Adverse Events (SAEs).
Description: The incidence of system and/or procedure related serious adverse events (SAEs) throughout the entire study period
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | The Reprieve System Implantation
Number analyzed (Participants) | 13
Participants | 1

2. Primary Outcome: Pain Assessment by Visual Analogue Scale (VAS) as Compared to Baseline at 6 Months Post Activation
Description: VAS score assessment at baseline and follow up visits was performed in two ways;
  1. Pain Diary VAS score- the analysis was based on the pain diary, processing the average daily VAS scores over seven consecutive days.
  2. Point VAS score- the analysis was based on the VAS score measurement recorded during the baseline visit and following 30 minutes stimulation at all follow up visits.Pain assessment by Visual Analogue Scale (VAS) as compared to baseline, post system activation.
  Visual Analogue Scale (VAS) for Pain Scores on a scale [0 - 10], higher values represent a worse outcome.
Time Frame: 1 Month, 3 Months, and 6 months post system activation
Population: Out of the 13 treated patients, one device was explanted approximately after 3 weeks of treatment. Thus, safety analysis is given for 13 patients and the performance analysis report on 12 patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Reprieve System Implantation
Number analyzed (Participants) | 12
score on a scale
  Pain Diary VAS Score - 1M post system activation | 3.94 (1.67)
  Pain Diary VAS score - 3M post system activation | 3.75 (1.67)
  Pain Diary VAS Score - 6M post system activation | 3.14 (1.52)
  Point VAS Score - 1M post system activation | 3.38 (2.48)
  Point VAS score - 3M post system activation | 2.79 (2.40)
  Point VAS Score - 6M post system activation | 2.42 (2.61)

3. Secondary Outcome: Clinical Success 6 Months Post Activation
Description: Clinical success at 6 months post activation was further assessed by:Short-form McGill pain questionnaire.
  McGill pain questionnaire Scores on a scale Range [0-60] points, higher values represent a worse outcome.
Time Frame: 1 Month, 3 Months, and 6 months post system activation
Population: Only 12 out of 13 patients completed the study. Thus, safety analysis is given for 13 patients and the performance analysis report on 12 patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The Reprieve System Implantation
Number analyzed (Participants) | 12
score on a scale
  McGill pain questionnaire - 1M post sys activation | 14 (12.1)
  McGill pain questionnaire - 3M post sys activation | 13.5 (13.4)
  McGill pain questionnaire - 6M post sys activation | 12.3 (14.3)

4. Secondary Outcome: Clinical Success 6 Months Post Activation
Description: Clinical success is defined as the effect of the BlueWind Reprieve System on the treatment of the following symptoms compared to baseline:
  - Pain related medication consumption/day
Time Frame: 6 months post activation
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | The Reprieve System Implantation
Number analyzed (Participants) | 12
Participants
  not consumed any pain related medication | 1
  didn't change medication consumption | 5
  Reduction in medication consumption | 6

5. Secondary Outcome: Clinical Success 6 Months Post Activation
Description: Clinical success was further assessed by: Quality of life questionnaire (SF-36 Health Survey) SF-36 Health Survey Scores on a scale [0 - 100], higher values represent a better outcome.
Time Frame: 1 Month, 3 Months, and 6 months post system activation
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | The Reprieve System Implantation
Number analyzed (Participants) | 12
score on a scale
  SF-36 Health Survey - 1M post system activation | 65.6 (5.2)
  SF-36 Health Survey - 3M post system activation | 66.4 (5)
  SF-36 Health Survey - 6M post system activation | 66.9 (4.2)

ADVERSE EVENTS:
Time Frame: 6 Month
Arm/Group | The Reprieve System Implantation
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 4/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Reprieve System Implantation (N=13)
low grade infection and delayed closure of surgical wound (Infections and infestations) | 1 (1) — The Reprieve implant was explanted approximately after 3 weeks of treatment.Patient was treated with antibiotics. The event terminated without further sequel and was classified as non-procedural related and its relationship to the device was unknown.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Reprieve System Implantation (N=13)
infection (Infections and infestations) | 2 (2)
implant site discolouration (General disorders) | 2 (2)
Skin irritatation (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Participating Institution and /or investigator may publish/present the results of the clinical investigation ("publication") only upon prior written consent provided by BlueWind Medical Ltd.